CLINICAL TRIAL: NCT04484675
Title: Comparative Study Between Inhaled and Intravenous Milrinone in Patients With Severe Pulmonary Hypertension Undergoing Cardiac Surgery
Brief Title: Inhaled and Intravenous Milrinone in Patients With Severe Pulmonary Hypertension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Mohamed EL -Asser,MD, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: milrinone in cardiadc surgery
Record Dates: First submitted 2020-07-13; First posted 2020-07-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Hypertension Due to Left Heart Disease
MeSH Terms: interventions — Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated randomization table divided patients into 2 equal groups randomly allocated patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group IH(inhaled milrinone) (Active Comparator): After induction of anesthesia and stable hemodynamics inhaled milrinone( 1 mg/ml) is initiated and intravenous placebo ( normal saline )infusion are administered
  Interventions: Drug: Milrinone inhalation
- Group Iv(Intravenous milrinone) (Active Comparator): After induction of anesthesia and stable hemodynamics inhaled placebo( normal saline) is initiated and intravenous ( 1 mg/ml) (0.5 μg/kg/min)infusion are administered
  Interventions: Drug: Milrinone infusion

INTERVENTIONS:
Drug: Milrinone inhalation — After induction of anesthesia and stable hemodynamics inhaled milrinone( 1 mg/ml) is initiated and intravenous placebo ( normal saline )infusion are administered
  Other Names: primacor
  Arms: Group IH(inhaled milrinone)
Drug: Milrinone infusion — After induction of anesthesia and stable hemodynamics inhaled placebo( normal saline) is initiated and intravenous ( 1 mg/ml) (0.5 μg/kg/min)infusion are administered
  Other Names: primacor
  Arms: Group Iv(Intravenous milrinone)

SUMMARY:
The investigator compared difference between inhaled and intravenous milirinone in patiens with severe pulmonary hypertension undergoing cardiac surgery

DETAILED DESCRIPTION:
Milrinone is widely used in cardiac surgery as an inotrope and pulmonary vasodilator agent But , intravenous milrinone has been associated with systemic hypotension and increased requirement for vasoactive drugs

The investigator compared difference between inhaled and intravenous milirinone in patiens with severe pulmonary hypertension undergoing cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo mitral valve surgery by cardiopulmonary bypass with estimated mean pulmonary artery pressure =>55 estimated by using preoperative Doppler echocardiography

Exclusion Criteria:

Patients were excluded if they had surgery without CPB, preoperative hemodynamic instability (deﬁned as acute requirement for vasoactive support or mechanical device),Patients with severe LV dysfunction (LV ejection fraction of less than 30% congenital heart disease, a contraindication to transesophageal echocardiography (TEE), emergency surgery or re-do surgeries severe renal or hepatic disease

, coagulopathy, and thromboembolic disease treated with anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
mean arterial pressure | change in mean arterial pressure is recorded 10 minutes after milrinone administration after induction (T1), at the end of nebulization (T2), before cardiopulmonary bypass (T3) and after cardiopulmonary bypass(T4)
  The effect of inhaled milrinone on mean arterial pressure is compared with the effect of intravenous milrinone

SECONDARY OUTCOMES:
mean pulmonary arterial pressure | change in mean pulmonary arterial pressure 10 minutes after milrinone administration
  The effect of inhaled milrinone on mean pulmonary pressure is compared with the effect of intravenous milrinone
systemic vascular resistance | change in systemic vascular resistance 10 minutes after milrinone administration
  The effect of inhaled milrinone on mean pulmonary pressure is compared with the effect of intravenous milrinone
pulmonary vascular resistance | change in pulmonary vascular resistance 10 minutes after milrinone administration
  The effect of inhaled milrinone on mean pulmonary pressure is compared with the effect of intravenous milrinone

CONTACTS AND LOCATIONS:
Overall Officials: Heba M EL-Asser, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denault AY, Bussieres JS, Arellano R, Finegan B, Gavra P, Haddad F, Nguyen AQN, Varin F, Fortier A, Levesque S, Shi Y, Elmi-Sarabi M, Tardif JC, Perrault LP, Lambert J. A multicentre randomized-controlled trial of inhaled milrinone in high-risk cardiac surgical patients. Can J Anaesth. 2016 Oct;63(10):1140-1153. doi: 10.1007/s12630-016-0709-8. Epub 2016 Jul 28. PMID 27470232
- [Background] Wang H, Gong M, Zhou B, Dai A. Comparison of inhaled and intravenous milrinone in patients with pulmonary hypertension undergoing mitral valve surgery. Adv Ther. 2009 Apr;26(4):462-8. doi: 10.1007/s12325-009-0019-4. Epub 2009 Apr 16. PMID 19381522